CLINICAL TRIAL: NCT01365286
Title: Heart Rate Lowering Efficacy and Respiratory Safety of Ivabradine in Patients With Obstructive Airway Disease
Brief Title: HR-lowering Efficacy and Respiratory Safety of Ivabradine in Patients With Obstructive Airway Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Lodz (Other)
Responsible Party: Sebastian Majewski, MD, Medical University of Lodz, Department of Pneumonology and Allergy
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Ivabradine2009-2011
Record Dates: First submitted 2011-05-31; First posted 2011-06-03 (Estimated); Last update posted 2012-06-12 (Estimated); Status verified 2011-05

CONDITIONS: Asthma, Chronic Obstructive Pulmonary Disease (COPD)
Keywords: asthma, chronic obstructive pulmonary disease, COPD, ivabradine, heart rate
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive | interventions — Ivabradine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ivabradine-Placebo (Active Comparator)
  Interventions: Drug: Ivabradine (Procoralan)
- Placebo-Ivabradine (Active Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ivabradine (Procoralan) — Ivabradine 7,5 mg b.i.d. for 5 days and Placebo b.i.d. for 5 days (Ivabradine-Placebo)
  Arms: Ivabradine-Placebo
Drug: Placebo — Placebo b.i.d. for 5 days and Ivabradine 7,5 mg b.i.d. for 5 days (Placebo-Ivabradine)
  Arms: Placebo-Ivabradine

SUMMARY:
The purpose of this study is to investigate heart rate lowering efficacy and respiratory safety of ivabradine in patients with asthma and COPD.

DETAILED DESCRIPTION:
In this double blind, placebo-controlled, crossover study, 20 asthmatics and 20 COPD patients received ivabradine 7,5 mg b.i.d. and placebo for 5 days in crossover manner. HR in ECG holter monitoring, peak expiratory flow rate (PEFR), symptoms, rescue medication consumption and AEs were evaluated in both periods of treatment.

ELIGIBILITY:
Inclusion Criteria:

* documented diagnosis of asthma or COPD in accordance with guidelines
* stable condition, defined as a disease without exacerbation for at least 1 month prior to study enrolment
* mean HR in holter ECG recording of ≥ 60 bpm

Exclusion Criteria:

* disease exacerbation in previous month
* inability to understand instructions on study procedures

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-05; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Heart rate | Change from baseline in heart rate during 5-day ivabradine and 5-day placebo treatment (24-hour ECG monitoring on the 3rd day)
  Difference in mean heart rate during ivabradine and placebo treatment

SECONDARY OUTCOMES:
Peak expiratory flow rate (PEFR) | Everyday measurement of morning and evening PEFR during 5-day ivabradine and 5-day placebo treatment
  Difference in mean daily PEFR during ivabradine and placebo treatment
Symptoms | Everyday symptom scoring during 5 day ivabradine and 5-day placebo treatment
  Difference in mean daily symptom score between ivabradine and placebo treatment
Rescue medication | Everyday rescue medication usage assessments during 5-day ivabradine and 5-day placebo treatment
  Difference in mean daily rescue medication use between ivabradine and placebo treatment
Number of participants with adverse events (AEs) | Number of patients with AEs evaluated throughout the study (5-day ivabradine and 5 day placebo treatment)
  Difference in number of participants with AEs between ivabradine and placebo treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Lodz, Department of Pneumonology and Allergy, Lodz, Poland

REFERENCES:
- [Background] Kannel WB, Kannel C, Paffenbarger RS Jr, Cupples LA. Heart rate and cardiovascular mortality: the Framingham Study. Am Heart J. 1987 Jun;113(6):1489-94. doi: 10.1016/0002-8703(87)90666-1. PMID 3591616
- [Background] Palatini P, Casiglia E, Pauletto P, Staessen J, Kaciroti N, Julius S. Relationship of tachycardia with high blood pressure and metabolic abnormalities: a study with mixture analysis in three populations. Hypertension. 1997 Nov;30(5):1267-73. doi: 10.1161/01.hyp.30.5.1267. PMID 9369286
- [Background] Hjalmarson A, Gilpin EA, Kjekshus J, Schieman G, Nicod P, Henning H, Ross J Jr. Influence of heart rate on mortality after acute myocardial infarction. Am J Cardiol. 1990 Mar 1;65(9):547-53. doi: 10.1016/0002-9149(90)91029-6. PMID 1968702
- [Background] Gillum RF, Makuc DM, Feldman JJ. Pulse rate, coronary heart disease, and death: the NHANES I Epidemiologic Follow-up Study. Am Heart J. 1991 Jan;121(1 Pt 1):172-7. doi: 10.1016/0002-8703(91)90970-s. PMID 1985358
- [Background] Fox K, Borer JS, Camm AJ, Danchin N, Ferrari R, Lopez Sendon JL, Steg PG, Tardif JC, Tavazzi L, Tendera M; Heart Rate Working Group. Resting heart rate in cardiovascular disease. J Am Coll Cardiol. 2007 Aug 28;50(9):823-30. doi: 10.1016/j.jacc.2007.04.079. Epub 2007 Aug 13. PMID 17719466
- [Background] Freemantle N, Cleland J, Young P, Mason J, Harrison J. beta Blockade after myocardial infarction: systematic review and meta regression analysis. BMJ. 1999 Jun 26;318(7200):1730-7. doi: 10.1136/bmj.318.7200.1730. PMID 10381708
- [Background] Frishman WH, Furberg CD, Friedewald WT. The use of beta-adrenergic blocking drugs in patients with myocardial infarction. Curr Probl Cardiol. 1984 Jun;9(3):1-50. doi: 10.1016/0146-2806(84)90015-x. No abstract available. PMID 6146495
- [Background] Gheorghiade M, Goldstein S. Beta-blockers in the post-myocardial infarction patient. Circulation. 2002 Jul 23;106(4):394-8. doi: 10.1161/01.cir.0000019582.39797.ef. No abstract available. PMID 12135934
- [Background] Farrell MH, Foody JM, Krumholz HM. beta-Blockers in heart failure: clinical applications. JAMA. 2002 Feb 20;287(7):890-7. doi: 10.1001/jama.287.7.890. PMID 11851583
- [Background] Fihn SD, Williams SV, Daley J, Gibbons RJ; American College of Cardiology; American Heart Association; American College of Physicians-American Society of Internal Medicine. Guidelines for the management of patients with chronic stable angina: treatment. Ann Intern Med. 2001 Oct 16;135(8 Pt 1):616-32. doi: 10.7326/0003-4819-135-8_part_1-200110160-00014. PMID 11601935
- [Background] Benson MK, Berrill WT, Cruickshank JM, Sterling GS. A comparison of four beta-adrenoceptor antagonists in patients with asthma. Br J Clin Pharmacol. 1978 May;5(5):415-9. doi: 10.1111/j.1365-2125.1978.tb01647.x. PMID 26371
- [Background] Schwartz S, Davies S, Juers JA. Life-threatening cold and exercise-induced asthma potentiated by administration of propranolol. Chest. 1980 Jul;78(1):100-1. doi: 10.1378/chest.78.1.100. PMID 7471827
- [Background] Williams IP, Millard FJ. Severe asthma after inadvertent ingestion of oxprenolol. Thorax. 1980 Feb;35(2):160. doi: 10.1136/thx.35.2.160. No abstract available. PMID 7376124
- [Background] Chang CL, Mills GD, McLachlan JD, Karalus NC, Hancox RJ. Cardio-selective and non-selective beta-blockers in chronic obstructive pulmonary disease: effects on bronchodilator response and exercise. Intern Med J. 2010 Mar;40(3):193-200. doi: 10.1111/j.1445-5994.2009.01943.x. Epub 2009 Mar 10. PMID 19383058
- [Background] DiFrancesco D, Camm JA. Heart rate lowering by specific and selective I(f) current inhibition with ivabradine: a new therapeutic perspective in cardiovascular disease. Drugs. 2004;64(16):1757-65. doi: 10.2165/00003495-200464160-00003. PMID 15301560
- [Background] Babu KS, Gadzik F, Holgate ST. Absence of respiratory effects with ivabradine in patients with asthma. Br J Clin Pharmacol. 2008 Jul;66(1):96-101. doi: 10.1111/j.1365-2125.2008.03160.x. Epub 2008 Mar 13. PMID 18341671
- [Background] Ageev FT, Makarova GV, Patrusheva IF, Orlova IaA. [The efficacy and safety of the combination of beta-blocker bisoprolol and if inhibitor I(f) ivabradine in patients with stable angina and chronic obstructive pulmonary disease]. Kardiologiia. 2010;50(10):22-6. Russian. PMID 21118175
- [Background] Masoli M, Fabian D, Holt S, Beasley R; Global Initiative for Asthma (GINA) Program. The global burden of asthma: executive summary of the GINA Dissemination Committee report. Allergy. 2004 May;59(5):469-78. doi: 10.1111/j.1398-9995.2004.00526.x. No abstract available. PMID 15080825
- [Background] Kjekshus JK. Importance of heart rate in determining beta-blocker efficacy in acute and long-term acute myocardial infarction intervention trials. Am J Cardiol. 1986 Apr 25;57(12):43F-49F. doi: 10.1016/0002-9149(86)90888-x. PMID 2871745
- [Background] Lechat P. Beta-blocker treatment in heart failure. Role of heart rate reduction. Basic Res Cardiol. 1998;93 Suppl 1:148-55. doi: 10.1007/s003950050243. PMID 9833143
- [Background] Fox K, Garcia MA, Ardissino D, Buszman P, Camici PG, Crea F, Daly C, De Backer G, Hjemdahl P, Lopez-Sendon J, Marco J, Morais J, Pepper J, Sechtem U, Simoons M, Thygesen K, Priori SG, Blanc JJ, Budaj A, Camm J, Dean V, Deckers J, Dickstein K, Lekakis J, McGregor K, Metra M, Morais J, Osterspey A, Tamargo J, Zamorano JL; Task Force on the Management of Stable Angina Pectoris of the European Society of Cardiology; ESC Committee for Practice Guidelines (CPG). Guidelines on the management of stable angina pectoris: executive summary: The Task Force on the Management of Stable Angina Pectoris of the European Society of Cardiology. Eur Heart J. 2006 Jun;27(11):1341-81. doi: 10.1093/eurheartj/ehl001. Epub 2006 May 30. No abstract available. PMID 16735367
- [Background] Ford ES, Giles WH, Croft JB. Prevalence of nonfatal coronary heart disease among American adults. Am Heart J. 2000 Mar;139(3):371-7. doi: 10.1016/s0002-8703(00)90076-0. PMID 10689247
- [Background] Lipworth BJ, Irvine NA, McDevitt DG. The effects of chronic dosing on the beta 1 and beta 2-adrenoceptor antagonism of betaxolol and atenolol. Eur J Clin Pharmacol. 1991;40(5):467-71. doi: 10.1007/BF00315224. PMID 1653143
- [Background] Lammers JW, Folgering HT, van Herwaarden CL. Respiratory tolerance of bisoprolol and metoprolol in asthmatic patients. J Cardiovasc Pharmacol. 1986;8 Suppl 11:S69-73. doi: 10.1097/00005344-198511001-00012. PMID 2439802
- [Background] Roche N, Huchon G. [Epidemiology of chronic obstructive pulmonary disease]. Rev Prat. 2004 Sep 15;54(13):1408-13. French. PMID 15497793
- [Background] Antonelli Incalzi R, Fuso L, De Rosa M, Forastiere F, Rapiti E, Nardecchia B, Pistelli R. Co-morbidity contributes to predict mortality of patients with chronic obstructive pulmonary disease. Eur Respir J. 1997 Dec;10(12):2794-800. doi: 10.1183/09031936.97.10122794. PMID 9493663
- [Background] Cazzola M, Calzetta L, Bettoncelli G, Novelli L, Cricelli C, Rogliani P. Asthma and comorbid medical illness. Eur Respir J. 2011 Jul;38(1):42-9. doi: 10.1183/09031936.00140310. Epub 2010 Dec 22. PMID 21177843
- [Background] Salpeter SR, Ormiston TM, Salpeter EE. Cardiovascular effects of beta-agonists in patients with asthma and COPD: a meta-analysis. Chest. 2004 Jun;125(6):2309-21. doi: 10.1378/chest.125.6.2309. PMID 15189956
- [Background] Sears MR. Adverse effects of beta-agonists. J Allergy Clin Immunol. 2002 Dec;110(6 Suppl):S322-8. doi: 10.1067/mai.2002.129966. PMID 12464943
- [Background] Fox K, Ford I, Steg PG, Tendera M, Ferrari R; BEAUTIFUL Investigators. Ivabradine for patients with stable coronary artery disease and left-ventricular systolic dysfunction (BEAUTIFUL): a randomised, double-blind, placebo-controlled trial. Lancet. 2008 Sep 6;372(9641):807-16. doi: 10.1016/S0140-6736(08)61170-8. Epub 2008 Aug 29. PMID 18757088
- [Background] Borer JS, Fox K, Jaillon P, Lerebours G; Ivabradine Investigators Group. Antianginal and antiischemic effects of ivabradine, an I(f) inhibitor, in stable angina: a randomized, double-blind, multicentered, placebo-controlled trial. Circulation. 2003 Feb 18;107(6):817-23. doi: 10.1161/01.cir.0000048143.25023.87. PMID 12591750
- [Background] Tardif JC, Ford I, Tendera M, Bourassa MG, Fox K; INITIATIVE Investigators. Efficacy of ivabradine, a new selective I(f) inhibitor, compared with atenolol in patients with chronic stable angina. Eur Heart J. 2005 Dec;26(23):2529-36. doi: 10.1093/eurheartj/ehi586. Epub 2005 Oct 7. PMID 16214830
- [Background] Kaneko A, Tachibana M. A voltage-clamp analysis of membrane currents in solitary bipolar cells dissociated from Carassius auratus. J Physiol. 1985 Jan;358:131-52. doi: 10.1113/jphysiol.1985.sp015544. PMID 2580078
- [Background] Demontis GC, Longoni B, Barcaro U, Cervetto L. Properties and functional roles of hyperpolarization-gated currents in guinea-pig retinal rods. J Physiol. 1999 Mar 15;515 ( Pt 3)(Pt 3):813-28. doi: 10.1111/j.1469-7793.1999.813ab.x. PMID 10066907
- [Background] Satoh TO, Yamada M. A bradycardiac agent ZD7288 blocks the hyperpolarization-activated current (I(h)) in retinal rod photoreceptors. Neuropharmacology. 2000 Apr 27;39(7):1284-91. doi: 10.1016/s0028-3908(99)00207-5. PMID 10760370
- [Derived] Majewski S, Slomka S, Zielinska-Wyderkiewicz E, Ciebiada M, Gorski P. Heart rate-lowering efficacy and respiratory safety of ivabradine in patients with obstructive airway disease: a randomized, double-blind, placebo-controlled, crossover study. Am J Cardiovasc Drugs. 2012 Jun 1;12(3):179-88. doi: 10.2165/11597400-000000000-00000. PMID 22409211